CLINICAL TRIAL: NCT04122560
Title: Fluconazole Pharmacokinetics, Including Bioavailability, in Obese Subjects After an Intravenous and Oral Administration (FOLIA)
Brief Title: Fluconazole Pharmacokinetics, Including Bioavailability, in Obese Subjects After an Intravenous and Oral Administration
Acronym: FOLIA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: St. Antonius Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UMCN-AKF-18.07
Record Dates: First submitted 2019-10-03; First posted 2019-10-10 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: Fluconazole; Candidiasis; Invasive Fungal Infections; Obesity
Keywords: fluconazole; candidiasis; invasive fungal infections; mycoses; antifungal agents
MeSH Terms: conditions — Candidiasis; Invasive Fungal Infections; Obesity; Mycoses | interventions — Fluconazole

STUDY DESIGN:
Intervention Model Description: Comparing a 2 groups of obese subjects vs 1 group of non-obese subjects
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Obese subjects (Experimental): Drug: Fluconazole tablet (diflucan) 200mg Single dose by oral administration of 400mg
  Drug: Fluconazole injection (diflucan) 400mg Single dose by intravenous infusion 400mg
  Interventions: Drug: Fluconazole 200mg tab; Drug: Fluconazole 2 MG/ML
- Non-obese subjects (Active Comparator): Drug: Fluconazole tablet (diflucan) 200mg Single dose by oral administration of 400mg
  Drug: Fluconazole injection (diflucan) 400mg Single dose by intravenous infusion 400mg
  Interventions: Drug: Fluconazole 200mg tab; Drug: Fluconazole 2 MG/ML

INTERVENTIONS:
Drug: Fluconazole 200mg tab — PO dose of 400mg
  Other Names: Diflucan
Drug: Fluconazole 2 MG/ML — IV dose of 400mg
  Other Names: Diflucan

SUMMARY:
The pharmacokinetics of fluconazole are expected to be different in obese patients compared to non-obese patients. The investigators will determine fluconazole and free fluconazole concentrations in 16 obese patients and 8 healthy volunteers, who will receive oral and intravenous fluconazole in a semi-simultaneous design.

A full pharmacokinetic curve will be obtained until 48 hours after intravenous administration.

DETAILED DESCRIPTION:
The pharmacokinetics of fluconazole are expected to be different in obese patients compared to non-obese patients. Therefore, extrapolation of data from healthy volunteers and is not possible.

To investigate these differences 16 obese patients and 8 healthy subjects will be studied.

Patients will receive fluconazole by semi-simultaneous design. Blood sampling for pharmacokinetic analysis will be retrieved through a central venous catheter. A maximum of 100 milliliter blood in total will be drawn for this study. Patients will be monitored daily during the treatment period for adverse events of the study drug.

Full pharmacokinetic curves will be taken after oral and intravenous administration. This pharmacokinetic analysis will enable the determination of bioavailability and enable the determination of intra-individual variability.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects BMI:

   1. obese groups: subject must have a BMI ≥35 kg/m2 at the time of inclusion or has undergone bariatric surgery;
   2. non-obese group: subject must have a BMI ≥18.5 and <30 kg/m2 at the time of inclusion;
2. Subject is at least 18 of age on the day of screening and not older than 65 years of age on the day of dosing;
3. Subject able and willing to sign the Informed Consent before screening evaluations.
4. If a woman, is neither pregnant nor able to become pregnant and is not nursing an infant.

   For the non-obese subjects the following additional inclusion criteria applies:
5. Subject is in good age-appropriate health condition as established by medical history, physical examination, electrocardiography, results of biochemistry and hematology within 6 weeks prior to study drug administration. Results of biochemistry and hematology should be within the laboratory's reference ranges (see Appendix A). If laboratory results are not within the reference ranges, the subject is included based on the investigator's judgment that the observed deviations are not clinically relevant. This should be clearly recorded.

Exclusion Criteria:

1. Documented history of sensitivity to fluconazole or similar azole-compound;
2. Documented history of the long QT syndrome (LQTS);
3. History of, or known abuse of drugs, alcohol or solvents (up until a maximum of three months before study drug administration);
4. Use of medication that has known relevant interaction with study drug as determined by the investigator up to 1 weeks prior to study drug administration;
5. Donation of blood or plasma to a blood bank or in a clinical study (except a screening visit) within 4 weeks prior to study drug administration;
6. Blood transfusion within 8 weeks prior to study drug administration;
7. Treatment with the concerning study drug up to 7 days before administration of the study drug;
8. Any other sound medical, psychiatric and/or social reason as determined by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-11-30 (Actual); Primary Completion 2021-03-23 (Actual); Study Completion 2021-03-23 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of fluconazole | 48 hours
  The concentration-time curve of fluconazole will be compared with that in non-obese subjects. Exposure is assessed by area-under-the-curve from zero to 48 hours (AUC0-48h)

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of fluconazole augmented dose | 48 hours
  The concentration-time curve of fluconazole will be compared with that in non-obese subjects. Exposure is assessed by area-under-the-curve from zero to 48 hours (AUC0-48h)

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - St. Antonius hospital, Nieuwegein
  - Radboudumc, Nijmegen

IPD SHARING:
Plan to Share IPD: No